CLINICAL TRIAL: NCT04412070
Title: A Pilot Study to Assess the Concordance of Genomic Alterations Between Urine and Tissue to Develop Precision Medicine-Based Immunotherapy Approaches in High-Risk NMIBC Patients
Brief Title: Assessement of the Concordance of Genomic Alterations Between Urine and Tissue in High-Risk NMIBC Patients
Acronym: ALU
Status: Terminated | Type: Observational
Why Stopped: The target enrollment was not reached at the end of recrutement period. The presence of a concurrent therapeutic clinical trial in the same department significantly limited patient availability for this study, making further recruitment not feasible.
Sponsor: Hopital Foch (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018_0087
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
Keywords: Muscle Invasive Bladder Cancer; Non-Muscle Invasive Bladder Cancer; cfDNA
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * One urine sample previously collected during patient's initial treatment and stored at the Biological Resources Center of Foch Hospital
  * Urine samples collected before each BCG (bacille Calmette Guerin) instillation
  * One blood sample collected before treatment with BCG during inclusion visit
  * One tumor sample previously collected during patient's initial treatment and stored in paraffin at the pathology department of Foch Hospital
  * One tumor sample collected in case of relapse during the 24 months follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with Non-Muscle invasive Bladder Cancer: Patients in this group will be enrolled before the start of their treatment with BCG. This will start within 4 weeks after the transurethral bladder resection, in accordance with the guidelines
- Patient with Muscle Invasive Bladder Cancer: Patients in this group will be enrolled in the study before surgical treatment by radical cystectomy

SUMMARY:
The analysis of cell-free tumor DNA (cfDNA) in plasma has emerged as a clinically relevant predictive and prognostic biomarker in several metastatic solid malignancies, and even now represents standard-of-care for prescription of some targeted therapies in non-small cell lung cancer (blood-based T790M companion diagnostic test). cfDNA can be detected not only in plasma but also in urine, even in patients with non-invasive disease. Recent studies found that the detection of genomic alterations in plasma of urothelial bladder carcinoma patients was relatively uninformative in the localized setting. However, urine cfDNA has been shown to provide a promising resource for robust whole-genome tumor profiling in clinically localized Muscle invasive Bladder cancer (MIBC) and Non-Muscle Invasive Bladder Cancer (NMIBC). Genomic alterations using a targeted next-generation sequencing (NGS) panel have been recently documented in a series of treatment-naïve high-risk NMIBC.

The investigator's aim is to determine whether liquid biopsies can be used as a new diagnostic assay to guide immunotherapeutic approaches in patients with high-risk NMIBC. The ultimate goal is to develop a "testing decision tree" to segment patients for informing on therapeutic decision and customizing treatment.

ELIGIBILITY:
Inclusion Criteria:

Common Inclusion Criteria

* Age ≥18 years at the time of screening.
* Capable of giving signed informed consent
* BCG-naïve (patients who have not received prior intravesical BCG or who previously received but stopped BCG more than 3 years before study entry are eligible).
* No prior radiotherapy to the bladder.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
* At screening, tumor tissue provision from the initial surgery, formalin-fixed and paraffin-embedded (FFPE) is mandatory for DNA extraction and next-generation sequencing.
* Absence of metastasis, as confirmed by a negative CT or MRI scan of the pelvis, abdomen and chest, no more than 4 weeks prior to the enrolment.
* Life expectancy of at least 12 weeks.
* Must be a candidate for BCG treatment.
* Adequate organ and marrow function as defined below:

Hemoglobin ≥9.0 g/dL Absolute neutrophil count ≥1.0 × 109/L Platelet count ≥75 × 109/L Serum bilirubin ≤1.5 × the upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.

Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN Measured creatinine clearance (CL) >40 mL/min or calculated creatinine CL >40 mL/min as determined by Cockcroft-Gault (using actual body weight) Males Creatinine CL = (Weight (kg) × (140 - Age))/(72 × serum creatinine (mg/dL)) (mL/min)

Females Creatinine CL = (Weight (kg) × (140 - Age) )/(72 × serum creatinine (mg/dL)) × 0.85 (mL/min) - Being covered by a national health insurance

Specific Inclusion Criteria for Non-Muscle Invasive Bladder Cancer (NMIBC) group

* Local histological confirmation (based on pathology report) of high-risk transitional cell carcinoma of the urothelium of the urinary bladder confined to the mucosa or submucosa (predominantly urothelial even though mixed histology are allowed). A high-risk tumor is defined as one of the following:
* T1 tumor
* High grade/G3 tumor
* CIS
* Multiple and recurrent and large (with diameter of largest evaluable node ≥3 cm) tumors (all conditions must be met in this point)
* Complete resection of all Ta/T1 papillary disease prior to enrolment, with the most recent TURBT (Trans Urethral Resection of Bladder Tumor) occurring 2 months or less prior to signing informed consent for this study. Patients with residual CIS after TURBT are eligible.
* At least one additional resection of the primary tumor has been performed in case of T1 tumors, or incomplete initial TURB, or in case of doubt about the completeness of a TURB, or if there is no muscle in the specimen (can be omitted if primary CIS (In situ cancer) only was found.)

Specific Inclusion Criteria for Muscle Invasive Bladder Cancer (MIBC) group Patients with histologically proven muscle-invasive bladder cancer (MIBC) scheduled before radical cystectomy.

Non-Inclusion Criteria:

Common Non-inclusion Criteria

* Evidence of lymphovascular invasion of bladder tumor, except if treatment with BCG is deemed to be the only clinically viable treatment (ie, clinical candidates of cystectomy and/or chemotherapy, etc are excluded).
* Known or documented absolute and/or relative contraindication of adjuvant intravesical BCG treatment.
* Concurrent extravesical (ie, urethra, ureter, or renal pelvis), non-muscle-invasive transitional cell carcinoma of the urothelium.
* Any concurrent chemotherapy, Intra Peritoneal, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
* Concurrent treatment with systemic immunostimulatory agents prior to the first dose of study treatment.
* History of allogenic organ transplantation. Patients with any history of allogenic stem cell transplantation are also excluded
* History of active primary immunodeficiency
* Pregnant or breastfeeding women
* Being deprived of liberty or under guardianship

Specific Non-inclusion Criteria for NMIBC group

- Evidence of muscle-invasive, locally advanced, metastatic, and/or extra-vesical bladder cancer (ie, T2, T3, T4, and / or stage IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population concerns :
  * Group 1 : patients with high-risk NMIBC treated by BCG therapy
  * Group 2 : patients with MIBC treated by radical cystectomy. This group will be considered as a positive control.
  During their conventional follow-up, a urine collection will be performed to each patient for testing of cell-free DNA. Genomic analysis of the primary tumor will be carried out on the tumor samples resetced during the initial diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Agreement rate between urine cell-free DNA and tumor tissue mutation profile | Day 0
  concordance rate between mutations identified in the tumor

SECONDARY OUTCOMES:
Prognostic value of Tumor Mutation Burden (TMB) | Day 0
  TMB will be calculated in the urine cell-free DNA for Each patient

CONTACTS AND LOCATIONS:
Overall Officials: Yanish Soorojebally, MD, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No